CLINICAL TRIAL: NCT03042039
Title: CareWell - Multi-level Integration for Patients With Complex Needs
Brief Title: Multi-level Integration for Patients With Complex Needs Facilitated by ICTs. A Shared Approach, Mutual Learning and Evaluation Are Expected to Create Synergies Among the Partners and to Bring Forward Integration of Care in Europe
Acronym: CAREWELL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Him SA (Other)
Responsible Party: Principal Investigator, Wouter A Keijser, General Manager of KRONIKGUNE, the Basque Centre for Health Services Research and Chronicity., Him SA
Other Study IDs: CareWell_EC_Grant No. 620983
Record Dates: First submitted 2017-01-24; First posted 2017-02-03 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Diabetes; Chronic Heart Failure; Frail Elderly Syndrome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group 'New Care': Frail elderly receiving care within new organisational models delivering integrated healthcare (IHC) supported by ICT infrastructure (electronically shared-care platform) as provided by pilot sites individually.
  Interventions: Other: New Care

INTERVENTIONS:
Other: New Care — New organisational care model delivering integrated healthcare (IHC) supported by ICT infrastructure (electronically shared-care platform).

SUMMARY:
CareWell will enable the delivery of integrated healthcare to frail elderly patients in a pilot setting through comprehensive multidisciplinary integrated care programmes where the role of ICTs can foster the coordination and patient centered delivery care. Carewell will focus in particular complex, multi-morbid elderly patients, who the patients most in need of health and social care resources (35% the total cost of Health Care System) and more complex interventions due to their frailty and comorbidities (health and social care coordination, monitoring, self-management of the patient and informal care giver). ICT platforms and communication channels that allow sharing information between healthcare and social care professionals involved in the delivery care of these patients, facilitating their coordination, increasing their resoluteness and avoiding duplicities when tackling patients´ diagnostic, therapeutic, rehabilitation or monitoring needs. Additionally, ICT-based platforms can improve the adherence to treatment, enhance self-care and increase patient awareness about their health status , as well as, improve the empowerment of informal caregivers, who usually take care of these patients.

According to this, it is hypothesized that the benefit of integrated care programmes based on (1) integrated care coordination and (2) patient empowerment & home support pathways supported by ICT is greater and essential for these patients. Care pathways will cut across organisational boundaries and will activate the most appropriate resources across the entire spectrum of healthcare and social care services available for both scheduled and emergency care. CareWell aims to scale up the services in pioneer regions and share their approach, learning from and supporting the other pilot sites which are at different levels of maturity in respect to designing, developing and implementing new ways of providing integrated care services.

DETAILED DESCRIPTION:
Frail elderly patients are characterised as having complex health and social care needs; they are at risk of hospital or residential care home admission, and require a range of high level interventions due to their frailty and multiple chronic conditions. A growing proportion of the population in OECD countries are age 65 and over: 15% in 2010, and expected to reach 22% by 2030. More than half of all older people have at least three chronic conditions, and a significant proportion have five or more.

A recent US study indicates that more than 95% of Medicare patients with a chronic disease such as congestive heart failure, depression, or diabetes have at least one other chronic condition, and the majority (80%, 71%, and 56%, respectively) have four or more chronic conditions. The CareWell project deals with multimorbid frail patients. Typically these patients have several diagnoses, the most frequent ones are:

* Chronic Obstructive Pulmonary Disease (COPD),
* Diabetes and
* Congestive Heart Failure (CHF).

The main objective of the CareWell study is to explore the data collection and analysis of health services' use. All sites are requested to upload their available data regarding service use, their flow chart on recruitment, and the demographic characteristics of end users. The evaluation has been conducted using the MAST multi-dimensional evaluation methodology adapted to the needs of CareWell project focusing on integrated healthcare.

MAST includes assessment of the outcomes of telemedicine applications divided into the following seven domains:

1. health problem and characteristics of the application;
2. safety;
3. clinical effectiveness;
4. patient perspectives;
5. economic aspects;
6. organisational aspects and
7. socio-cultural, ethical and legal aspects. Each domain will be addressed and studied through a range of methodological approaches, quantitative, qualitative and modelling.

Patients distributed in six sites will be recruited and assessed at baseline and be followed up during a period of six months. Data is to be collected from different sources, including administrative databases, questionnaires and personal interviews.

All 6 CareWell sites are to conduct cohort studies, which means that a group of people with similar characteristics are followed over a period of time. Potential participants are selected by screening electronic healthcare records and/or the hospital / national databases and/or during long term condition annual reviews in the community setting.

Candidates are informed about the nature and the objectives of the evaluation. Once candidates have signed the informed consent form, if necessary, they participate in the evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years.
2. Presence of at least two chronic diseases included in the Charlson Comorbidity Index (CCI) [4]. At least one of the comorbid conditions must be one of the following conditions: Chronic obstructive pulmonary disease (COPD), diabetes mellitus (both insulin-dependent and noninsulin-dependent) or chronic heart failure (CHF).
3. Fulfilling local/national/organisational criteria of frailty: increased vulnerability, complex health needs, and at high risk of hospital or care home admission.
4. Participants have to be able to understand and to comply with study instructions and requirement, either independently or with help from a carer.

Exclusion Criteria:

1. Subjects who have either been registered with an active cancer diagnosis under treatment, have undergone an organ transplant, or are undergoing dialysis prior to enrolment.
2. Subjects who are candidates for palliative care (with life expectancy less than one year, clinically evaluated).
3. People with an AIDS diagnosis.
4. People living in care homes where their daily health, care and wellbeing needs are met by staff (nurses and support staff) employed within the home.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Frail elderly living in one of the 6 CareWell sites
Sampling Method: Probability Sample
Enrollment: 1712 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Total number of hospital admissions per participant measured at end of study (at approx 12 months) | Total of hospital admissions as measured after (approximately) 12 months (= end of study)
  The total of (planned and unplanned) hospital admissions

SECONDARY OUTCOMES:
Change in generic health related/functional quality of life (1) by assessing Charlson Comorbidity Index (CCI) | Change in CCI between baseline and after (approximately) 12 months (=end of study)
  Charlson Comorbidity Index (CCI)
Change in Generic health related/functional quality of life (2) by assessing Barthel index | Change in Generic health related/functional quality of life as assessed based on BARTHEL INDEX scores between baseline and (approximately) after 12 months (=end of study)
  Barthel index
Change in Psychological measures (1) by assessing Geriatric Depression Scale | Changes in Psychological measures as assessed based on GDS-SF between baseline, midterm (after approximately 6 months) and after (approximately) 12 months (=end of study)
  Geriatric Depression Scale (GDS Short Form)
Change in Psychological measures (2) by measuring Hospital Anxiety and Depression Scale | Changes in Psychological measures as assessed based on HADS measurements between baseline, midterm (after approximately 6 months) and after (approximately) 12 months (=end of study)
  Hospital Anxiety and Depression Scale (HADS Scale)
Changes in the User perspectives (1) by measuring PIRU questionnaire on user experience of Integrated Care (IC) by measuring Policy Research Unit in Policy Innovation Research questionnaire | Changes in User perspectives as assessed based on PIRU scores between baseline, midterm (after approximately 6 months) and after (approximately) 12 months (=end of study)
  Policy Research Unit in Policy Innovation Research (PIRU) questionnaire on user experience of Integrated Care (IC)
Changes in User perspectives (3) by measuring Carer perspectives of integration according to eCCIS | Changes in User perspectives as assessed based on eCCIS measurements of CARERS between baseline, midterm (after approximately 6 months) and after (approximately) 12 months (=end of study)
  Carer perspectives of integration according to eCCIS
Changes in User perspectives (4) by measurement of NHS LTC6 Questionnaire | Changes in NHS-LTC6 measurements between baseline, midterm (after approximately 6 months) and after (approximately) 12 months (=end of study)
  National Health Services (NHS) LTC6 Questionnaire
Economic aspects (1) as measured based on the total of Efforts related to service development & implementation during the study (between start and 12 months) | Economic aspects as assessed based on measurements of total efforts related to Development and Implementation of Services during the period between baseline and after (approximately) 12 months (=end of study)
  Efforts related to service development & implementation
Changes in Economic aspects (2) as measured based on the total of Efforts related to service during the operation or use of the study (between starts and 12 months) | Economic aspects as assessed based on measurements of total efforts related to Service Operations during the period between baseline and after (approximately) 12 months (=end of study)
  Efforts related to service operation or use
Changes in Economic aspects (3) as measured based on the total of Equipment costs during the project, between start and after 12 months | Economic aspects as assessed based on measurements of total of Costs of Equipment during the period between baseline and after (approximately) 12 months (=end of study)
  Equipment costs
Changes in Economic aspects (4) based on measurements of Service effectiveness benefits during study (between start and 12 months) | Total of Benefits in Effectiveness of Services during the period between baseline and after (approximately) 12 months (=end of study)
  Service effectiveness benefits
Changes in of Economic aspects (5) based on measurements of Service efficiency benefits during study (between start and 12 months) | Economic aspects as assessed based on measurements of total of Benefits in Efficiency of Services during the period between baseline and after (approximately) 12 months (=end of study)
  Service efficiency benefits
Changes in Economic aspects (6) based on changes in measurements Changes Willingness to pay between start en end of study (12 months) | Economic aspects as assessed based on measurements of Changes in Willingness To Pay for Services between baseline and after (approximately) 12 months (=end of study)
  Changes Willingness to pay
Impact on Organisational aspects (1) as measured with impact on staff between start and study end (after 12 months) | Total of Services' Impact On Staff during the period between baseline after (approximately) 12 months (=end of study)
  Impacts on staff
Impact on Organisational aspects (2) as measured with impact on involved organisations between start study and end (12 months) | Total of Services' Impact On Organisations during the period between baseline and after (approximately) 12 months (=end of study)
  Impacts on organisation
Changes in Overall service effectiveness and specific outcome measures (1) as measured with Admission-Discharge Duration of admissions between start and study end | Changes in Overall service effectiveness and specific outcome assessed based on change between Average of Duration of each Admission throughout study between baseline and after (approximately) 12 months (=end of study)
  Admission-Discharge Duration
Changes in Overall service effectiveness and specific outcome measures (2) as measured with Indication for hospitalisation of all admissions between start and study end (12 months) | Changes in Overall service effectiveness and specific outcome by recording of Admission Indication throughout study between baseline and after (approximately) 12 months (=end of study)
  Indication for hospitalisation
Changes in Overall service effectiveness and specific outcome measures (3) as measured with Re-hospitalisation rates within 30 days after dismissal between start and end study (12 months) | Changes in Overall service effectiveness and specific outcome as assessed based on change between measurements of total of re-hospitalization within 30 days after last admission throughout study between baseline and after (approx.) 12 months (=study end)
  Re-hospitalisation within 30 days
Change in Overall service effectiveness and specific outcome measures (4) as assessed with Origin before Admission of all admissions between start and end of study (12 months) | Changes in Overall service effectiveness and specific outcome by recording of Origin ad each Admission throughout study between baseline and after (approximately) 12 months (=end of study)
  Origin before Admission
Change in Overall service effectiveness and specific outcome measures (5) as assessed with Discharge destiny of all discharges between start and end of study (12 months) | Changes in Overall service effectiveness and specific outcome by recording of Destiny after each discharge throughout study between baseline and end of study (12 months)
  Discharge destiny
Change in Disease specific health status measurement (1) as measured with HbA1c of diabetes patients between start and end of study (12 months) | Changes in Disease specific health status based on measurements of HbA1c between baseline and after (approximately) 12 months (=end of study)
  HbA1c
Change in Disease specific health status measurement (2) as measured with blood glucose levels of all diabetes patients between start and end of study (12 months) | Changes in Disease specific health status based on measurements of Blood Glucose between baseline and after (approximately) 12 months (=end of study)
  Blood glucose
Change in Disease specific health status measurement (3) as measured with heart rate measurements of all chronic heart failure patients between start and study end (12 months) | Changes in Disease specific health status based on measurements of Heart Rate between baseline and after (approximately) 12 months (=end of study)
  Heart rate
Change in Disease specific health status measurement (4) as measured with blood pressure of all patients with chronic heart failure between start and end of study (12 months) | Changes in Disease specific health status based on measurements of blood Pressure between baseline and after (approximately) 12 months (=end of study)
  Blood pressure
Change of Disease specific health status measurement (5) as measured with weight of all patients with chronic heart failure between start and end of study (12 months) | Changes in Disease specific health status based on measurements of Weight between baseline and after (approximately) 12 months (=end of study)
  Weight
Change in Disease specific health status measurement (6) as measured with BMI of all patients with chronic heart failure between start and end of study (12 months) | Changes in BMI between baseline and after (approximately) 12 months (=end of study)
  BMI

CONTACTS AND LOCATIONS:
Locations (5):
- Higher or Secondary Education Establishments, Zagreb, Croatia
- Agenzia Regionale Sanitaria Pugliese, Bari, Italy
- Urzad Marszalkowski Wojewodztwa Dolnoslaskiego, Wroclaw, Poland
- Servicio Vasco de Salud Osakidetza, Vitoria-Gasteiz, Spain
- Bronllys Hospital, Bronllys, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kidholm K, Ekeland AG, Jensen LK, Rasmussen J, Pedersen CD, Bowes A, Flottorp SA, Bech M. A model for assessment of telemedicine applications: mast. Int J Technol Assess Health Care. 2012 Jan;28(1):44-51. doi: 10.1017/S0266462311000638. PMID 22617736
- [Background] Agha Z, Schapira RM, Maker AH. Cost effectiveness of telemedicine for the delivery of outpatient pulmonary care to a rural population. Telemed J E Health. 2002 Fall;8(3):281-91. doi: 10.1089/15305620260353171. PMID 12419022
- [Background] Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, Oxman AD, Moher D; CONSORT group; Pragmatic Trials in Healthcare (Practihc) group. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008 Nov 11;337:a2390. doi: 10.1136/bmj.a2390. PMID 19001484
- [Background] Kopec JA, Fines P, Manuel DG, Buckeridge DL, Flanagan WM, Oderkirk J, Abrahamowicz M, Harper S, Sharif B, Okhmatovskaia A, Sayre EC, Rahman MM, Wolfson MC. Validation of population-based disease simulation models: a review of concepts and methods. BMC Public Health. 2010 Nov 18;10:710. doi: 10.1186/1471-2458-10-710. PMID 21087466
- [Background] Speroff T, O'Connor GT. Study designs for PDSA quality improvement research. Qual Manag Health Care. 2004 Jan-Mar;13(1):17-32. doi: 10.1097/00019514-200401000-00002. PMID 14976904
- [Background] Hiligsmann M, Gathon HJ, Bruyere O, Ethgen O, Rabenda V, Reginster JY. Cost-effectiveness of osteoporosis screening followed by treatment: the impact of medication adherence. Value Health. 2010 Jun-Jul;13(4):394-401. doi: 10.1111/j.1524-4733.2009.00687.x. Epub 2010 Jan 21. PMID 20102558
- [Background] Lega F, DePietro C. Converging patterns in hospital organization: beyond the professional bureaucracy. Health Policy. 2005 Nov;74(3):261-81. doi: 10.1016/j.healthpol.2005.01.010. PMID 16226138
- [Derived] Mateo-Abad M, Gonzalez N, Fullaondo A, Merino M, Azkargorta L, Gine A, Verdoy D, Vergara I, de Manuel Keenoy E. Impact of the CareWell integrated care model for older patients with multimorbidity: a quasi-experimental controlled study in the Basque Country. BMC Health Serv Res. 2020 Jul 3;20(1):613. doi: 10.1186/s12913-020-05473-2. PMID 32620116
- See also: Project Website CareWell — http://carewell-project.eu/norm/home.html